CLINICAL TRIAL: NCT06187948
Title: An Informative Video Before Planned External Cephalic Version - Does it Reduce Maternal Anxiety and Improve Chances of Success? - a Randomized Control Trial
Brief Title: An Informative Video Before Planned External Cephalic Version
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0214-22
Record Dates: First submitted 2023-05-02; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-04

CONDITIONS: Breech Presentation
Keywords: breech presentation; external cephalic version; maternal anxiety; informative video
MeSH Terms: conditions — Breech Presentation | interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1. group that watches an informative video (Experimental): All participants in the intervention group watches an informative video on recruitment. This video describes in detail the expected external cephalic version process.
  Interventions: Other: Video
- 2. group that does not watch an informative video (No Intervention): this group do not watch an informative video before recruitment

INTERVENTIONS:
Other: Video — All participants in the intervention group watches an informative video on recruitment. This video describes in detail the expected external cephalic version process.
  Arms: 1. group that watches an informative video

SUMMARY:
A randomized control trial to investigate whether an informative video before planned external cephalic version reduces maternal anxiety and improves chances of success.

DETAILED DESCRIPTION:
Women with a breech presentation scheduled to undergo an external cephalic version that meet the criteria are recruited in the Emergency Room by offering every woman that is scheduled to undergo an external cephalic version to participate. Women who agree to participate are asked to sign an inform consent, and are randomized to intervention group and control group. In the Emergency Room sonographic data is collected including amniotic fluid index, engaged presenting part, sonographic and clinical estimation of fetal weight, place of the placenta and various angles between the fetus and the bladder (These data are collected for the study). All participants in the intervention group watches an informative video on recruitment. This video describes in detail the expected external cephalic version process.

Before the external cephalic version and an hour after a successful or an unsuccessful external cephalic version the situation-specific anxiety is measured using the State-Trait Anxiety Inventory score (Attached).

ELIGIBILITY:
Inclusion Criteria:

* Women between ages 18-45
* with a singleton gestation
* at gestational week of 36 weeks 0 days until 38 weeks 0 days
* who admitted labor word for external cephalic version .

Exclusion Criteria:

* Women who had a past cesarean section
* Women with oligohydramnios (Amniotic fluid index < 5 cm)
* Women who had a past external cephalic version
* Women with a failed external cephalic version in current pregnancy
* Women who take medication for depression/anxiety disorders
* Women with a complicated pregnancy including fetal anomalies, polyhydramnios…

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnancy
Enrollment: 200 (Estimated)
Dates: Start 2023-12-26 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
higher success rates. | 4 years
  Comparing the percentage of successful External Cephalic Version (ECV) procedures between patients who watched an informative video about the procedure and those who did not receive this intervention.

SECONDARY OUTCOMES:
impact of watching an informative video before external cephalic version on maternal anxiety levels | 4 years
  Assessing anxiety levels using the State-Trait Anxiety Inventory, administered at two time frames - before the External Cephalic Version (ECV) and an hour after - to determine if women who watch an informative video about the procedure experience lower anxiety compared to those who do not.

CONTACTS AND LOCATIONS:
Overall Officials: Dorit Ravid, Dr, Study Director — Meir Hospital
Locations (1):
- Meir Medical Center, Kfar Saba, Israel